CLINICAL TRIAL: NCT05675722
Title: Phase 1 Trial Of Implantation Of Vaginal Construct For Patients With Vaginal Aplasia
Brief Title: Implantation Of Vaginal Construct For Patients With Vaginal Aplasia
Acronym: TEV
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00091486
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Congenital Mullerian Duct Anomaly
Keywords: Vaginal Abnormality

STUDY DESIGN:
Intervention Model Description: Ten women, ages 15-45 years, meeting criteria will undergo vaginal/vulva biopsy and biologic vaginal-construct implantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- autologous vaginal construct for patients with vaginal aplasia (Experimental): Biologic vaginal construct, surgically implanted into native vaginal site
  Interventions: Biological: biologic vaginal-construct implantation

INTERVENTIONS:
Biological: biologic vaginal-construct implantation — biologic Tissue Engineered Vagina (TEV), which provides an epithelial layer for the luminal aspect and a smooth muscle layer for protecting the openness of the hollow tube, mimicking the cellular orientation and architecture of the vagina. Autologous cells isolated from vagina/vulva remnants offset any potential for immunological rejection.

SUMMARY:
In this Phase 1, single site, clinical trial, Vulvar/vaginal Smooth muscle cells (SMC) and Epithelial Cells (EPC) are isolated from autologous patient's biopsy

DETAILED DESCRIPTION:
The cells are expanded in vitro and seeded on scaffold and matured - The final Tissue Engineered Vagina (TEV) is implanted into the native vaginal site

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital Mullerian duct anomaly that includes absence or obliteration of all or part of the vagina, as confirmed on pelvic MRI
* Females between the ages of 15 and 45 years
* Patients with stable medical comorbidities
* Patients that are willing to comply with all study instructions and are willing to return for study follow-up visits

Exclusion Criteria:

* Patients with a history of surgery in the target area more recent than the last 6 months
* Patients with an active vaginal area infection or urinary infection as evidenced by clinical exam or culture result
* Patients with a history of keloid scarring
* Patients who are currently taking anti-platelet medications or blood thinners
* Patients with a history of clotting disorder
* Patients with autoimmune disease or immune disorder
* Patients requiring concomitant use of or treatment with immunosuppressive agents
* Patients with a history of systemic conditions, including but not limited to HIV, thrombocytopenia, uncontrolled diabetes and chronic liver disease (including Hepatitis B or C), that the Investigator believes may jeopardize the safety of the patient to participate in the study
* Patients with evidence or diagnosis of any primary coagulation disorder (including concomitant anticoagulation therapy at enrollment)
* Patients who have been treated with any other investigational drug or participated in any investigational study within 30 days prior to enrollment in this study
* Patients with neurological disorders (e.g., multiple sclerosis, Parkinson's disease)
* Patients who are current tobacco users
* Patients with alcohol/drug abuse problems
* Patients with any systemic disease
* Patients with any psychiatric disorders
* Inability to participate in all necessary study activities due to physical or mental limitations.
* Any circumstance in which the investigator deems participation in the study is not in the subject's best interest
* The following vital sign cut-off values, laboratory cut-off values and ECG reading will be monitored as the exclusion criteria in the biopsy visit and again before the implantation surgery BP systolic >160 or <90 millimeters of mercury (mmHg) or diastolic >100 or<60 millimeters of mercury (mmHg) Pulse <60 or >105bpm Respiratory Rate < 9 and >20 Temp > 100.4 degrees Fahrenheit Liver enzymes >2 times the upper limit of normal (ULN) Abnormal bilirubin unless subject has Gilbert's glomerular filtration rate (eGFR) < 60 mL/min/ 1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) HbA1C > 8% Hb <10 mg/dL Platelet Count <100,000 O2 saturation <95%
* If a vital sign or lab value results in exclusion, the subject could be rescreened later

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — a diagnosis of vaginal agenesis due to a Mullerian duct anomaly
Enrollment: 10 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Serious Adverse Events | Month 36
  bleeding, pain, visceral injury, vaginal scarring, contraction, or infection
Quality of Life Scores | Baseline
  The Quality of Life Scores (QOLS) is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112 - the higher score indicates the higher quality of life
Quality of Life Scores | Month 36
  The Quality of Life Scores (QOLS) is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112 - the higher score indicates the higher quality of life

SECONDARY OUTCOMES:
Change in Quality of life Female Sexual Function Index (FSFI) Scores | Month 3, Month 6, Month 12, and Month 36
  The Female Sexual Function Index (FSFI) is a multidimensional measure of female sexual functioning with 19 items that have ordinal, Likert- type response formats and are scored from 0 (or 1) to 5. The scoring algorithm sums items on each domain/sub-scale and then scales the sums so that each subscale has a maximum score of 6 - The FSFI is a survey measuring the sexual functioning of women in six different domains: desire, arousal, lubrication, orgasm, satisfaction and pain - Higher scores indicate better functioning

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Matthews, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No